CLINICAL TRIAL: NCT02281149
Title: Adjuvant Radiotherapy in Breast With Intensity Modulated by Tomotherapy: Evaluation of the Toxicity and Quality of Life
Brief Title: Adjuvant Radiotherapy in Breast With Intensity Modulated by Tomotherapy:
Acronym: TOMOBREAST
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: TOMOBREAST-1307
Record Dates: First submitted 2014-10-28; First posted 2014-11-03 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiotherapy; intensity modulation; toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Adjuvant radiotherapy after lumpectomy allows a local long-term control of the order 85 to 95% with a survival rate equivalent to that of the totally mastectomy. The diminution of the local recurrence rate after irradiation post- lumpectomy is also associated to a best global survival than only the surgery. The adjuvant radiotherapy after partially or totally mastectomy for the progressive tumors is a therapeutic standard (Early Breast Cancer Trialists' Collaborative Group 2011). The aim of our trial of routine care is to record our practices under this breast adjuvant radiotherapy.

DETAILED DESCRIPTION:
Patients responding criteria for selection and not objecting to participate in this trial will address the quality of life questionnaires at baseline and during their standard follow-up (1, 6, 12 and 24 months after the end of radiotherapy). The data of toxicity and disease-free survival will be collected from data on medical record of the patient.

The therapeutic support and monitoring are standard.

ELIGIBILITY:
Inclusion Criteria:

1-Patient with breast cancer proved by histology and treated surgically 2. Relevant of adjuvant radiotherapy after partial or total mastectomy with or without lymph node irradiation 3- Age ≥ 18 years 4- Information and no opposition to the patient

Exclusion Criteria:

1. - Metastatic disease
2. - Patient having another severe disease or uncontrolled which could jeopardize the trial participation
3. - pregnant or breastfeeding woman 4-inability to do follow-up medical care of clinical trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective study of routine care done on women with breast cancer treated by adjuvant radiotherapy with intensity modulated
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
acute and tardive toxicity according to NCI-CTCAE v4.0 | up to 5 years
  according to NCI-CTCAE v4.0

SECONDARY OUTCOMES:
Quality of life according to QLQC-30 | up to 24 months
  Quality of life according to QLQC-30
Quality of life according to BR-23 module | up to 24 months
  Quality of life according to BR-23 module
Disease free survival | up to 5 years
  according to RECIST 1.1
esthetic results | up to 5 years
  by physician and patient according to a scale (good, excellent, moderate and poor)

CONTACTS AND LOCATIONS:
Overall Officials: David PASQUIER, MD, Principal Investigator — Centre Oscar Lambret
Locations (2):
- France (2):
  - Centre Léonard de Vinci, Douai
  - Centre Oscar Lambret, Lille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquier D, Bataille B, Le Tinier F, Bennadji R, Langin H, Escande A, Tresch E, Darloy F, Carlier D, Crop F, Lartigau E. Correlation between toxicity and dosimetric parameters for adjuvant intensity modulated radiation therapy of breast cancer: a prospective study. Sci Rep. 2021 Feb 11;11(1):3626. doi: 10.1038/s41598-021-83159-3. PMID 33574446